CLINICAL TRIAL: NCT06882785
Title: A Phase 3, Randomized, Two-part Study With a 5-week Double-blind Part (Randomized, Parallelgroup, Placebo-controlled) Followed by a 52-week Open-label Extension Part to Evaluate the Efficacy and Safety of KarXT in Acutely Psychotic Japanese Adult Patients With Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5) Schizophrenia
Brief Title: A Study to Evaluate the Efficacy and Safety of KarXT in Acutely Psychotic Japanese Adult Participants With Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN012-0019
Record Dates: First submitted 2025-03-17; First posted 2025-03-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Administration of KarXT (Active Comparator)
  Interventions: Drug: KarXT
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510
  Arms: Administration of KarXT
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KarXT in acutely psychotic Japanese adult participants with schizophrenia

ELIGIBILITY:
Inclusion Criteria

* Participants must have a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the Diagnostic and Statistical Manual of Mental Disorders⎯Fifth Edition (DSM-5) criteria and confirmed by Mini International Neuropsychiatric Interview (MINI).
* Participants must have a PANSS total score between 80 and 120, inclusive.
* Participants must have a CGI-S score of ≥ 4.

Exclusion Criteria

* Participants must not have any primary DSM-5 disorder other than schizophrenia within 12 months before screening.
* Participants must not be newly diagnosed or experiencing their first treated episode of schizophrenia.
* Participants must not have any history or presence of clinically significant medical conditions.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-09-23 (Estimated); Study Completion 2029-08-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | At week 5
  Double-Blind Part
Number of participants with treatment-emergent adverse events (TEAEs) | At Week 52 from OLE baseline
  Open-label extension (OLE) Part

SECONDARY OUTCOMES:
Change from baseline in PANSS positive score | At week 5
  Double-blind Part
Change from baseline in PANSS negative score | At week 5
  Double-blind Part
Change from baseline in PANSS Negative Marder Factor score | At week 5
  Double-blind Part
Change from baseline in Clinical Global Impressions-Severity (CGI-S) score | At week 5
  Double-blind Part
The percentage of PANSS responders (a ≥ 30% change in PANSS total score) | At week 5
  Double-blind Part
Number of participants wtih adverse events (AEs) | Up to day 35
  Double-blind Part
Number of participants wtih adverse events of special interest (AESIs) | Up to week 57
Number of participants with procholinergic symptoms | Up to week 57
Number of participants with anticholinergic symptoms | Up to week 57
Change from baseline in Simpson-Angus Scale (SAS) score | Up to day 35
  Double-blind Part
Change from baseline in Barnes Akathisia Rating Scale (BARS) score | Up to day 35
  Double-blind Part
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) score | Up to day 35
  Double-blind Part
Change from baseline in body weight | Up to day 35
  Double-blind Part
Change from baseline in body mass index (BMI) | Up to day 35
  Double-blind Part
Blood pressure (BP) sitting and standing after 2 minutes | Up to week 57
Heart rate (HR) sitting and standing after 2 minutes | Up to week 57
Number of participants wtih a change from baseline in hematology evaluations | Up to week 57
Number of participants wtih a change from baseline in clinical chemistry evaluations | Up to week 57
Number of participants wtih a change from baseline in coagulation evaluations | Up to week 57
Number of participants wtih a change from baseline in urinalysis evaluations | Up to week 57
Number of participants wtih a change from baseline in drug screen evaluations | Up to week 57
Number of participants wtih a change from baseline in 12-lead electrocardiogram (ECG) evaluations | Up to week 57
Number of participants wtih physical examination abnormalities | Up to week 57
Number of participants wtih suicidal ideation with the use of the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to week 57
International Prostate Symptom Score (IPSS) | Up to week 57
  Male participants ≥ 45 years of age only
Area under the plasma concentration-time curve (AUC) | Up to day 35
  Double-blind Part
Maximum observed plasma concentration (Cmax) | Up to day 35
  Double-blind Part
Time of maximum observed plasma concentration (Tmax) | Up to day 35
  Double-blind Part
Number of participants wtih serious TEAEs | Up to week 57
  OLE Part
Number of participants wtih TEAEs leading to discontinuation of study intervention | Up to week 57
  OLE Part
Change from OLE baseline in PANSS total score | At week 57
  OLE Part
Change from OLE baseline in CGI-S score | At week 57
  OLE Part
Percentage of PANSS responders | At week 57
  OLE Part

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (55):
- Japan (55):
  - Hotei Hospital, Kōnan, Aichi-ken
  - Local Institution - 0056, Nagoya, Aichi-ken
  - Okehazama Hospital, Toyoake, Aichi-ken
  - Fujita Health University, Toyoake, Aichi-ken
  - National Kohnodai Medical Center., Ichikawa, Chiba
  - National Hospital Organization Shimofusa Psychiatric Medical Center, MIdori-ku, Chiba-shi, Chiba
  - Local Institution - 0032, Iizuka, Fukuoka
  - Local Institution - 0037, Kitakyushu, Fukuoka
  - Shiranui Hospital, Omuta, Fukuoka
  - Takeda General Hospital - Aizuwakamatsu, Aizu-Wakamatsu, Fukushima
  - Local Institution - 0044, Toki, Gifu
  - Kure Medical Center, Kure, Hiroshima
  - Goryokai Medical Corporation - Goryokai Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Local Institution - 0025, Hadano-shi, Kanagawa
  - Fujimidai Hospital, Hiratsuka, Kanagawa
  - Local Institution - 0052, Sagamihara, Kanagawa
  - Tsurumi Nishii Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Hino Hospital - Yokohama, Yokohama, Kanagawa
  - Yuge Hospital, Kumamoto, Kumamoto
  - Local Institution - 0019, Yatsushiro, Kumamoto
  - National Hospital Organization Maizuru Medical Center, Maizuru, Kyoto
  - Miyakonojo Shinsei Hospital, Miyakonojō, Miyazaki
  - Local Institution - 0014, Komoro, Nagano
  - Local Institution - 0050, Matsumoto, Nagano
  - Local Institution - 0051, Ginowan, Okinawa
  - Osaka Psychiatric Medical Center, Hirakata, Osaka
  - Kansai Medical University Medical Center, Moriguchi, Osaka
  - Nagaokai Medical Corporation - Neyagawa Sanatorium, Neyagawa, Osaka
  - Shin-Abuyama Hospital, Takatsuki, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Rainbow and Sea Hospital, Karatsu-shi, Saga-ken
  - Inuo Hospital, Tosu, Saga-ken
  - Saitama Konan Hospital, Kumagaya, Saitama
  - Dokkyo Medical University Hospital, Shimotsuga, Tochigi
  - Local Institution - 0043, Utsunomiya, Tochigi
  - Local Institution - 0012, Hachiōji, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Asuka Hospital, Machida, Tokyo
  - Local Institution - 0053, Ōta-ku, Tokyo
  - Tokyo Metropolitan Matsuzawa Hospital, Setagaya City, Tokyo
  - Narimasu Kosei Hospital, tabashi City, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Kuramitsu Hospital, Fukuoka
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki
  - Local Institution - 0055, Okayama
  - Local Institution - 0018, Okinawa
  - Local Institution - 0031, Osaka
  - Saitama Neuropsychitric Institute, Saitama
  - Local Institution - 0039, Tokushima
  - Local Institution - 0033, Tottori
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata Sakuracho Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html